CLINICAL TRIAL: NCT01287754
Title: A Study of Erlotinib (Tarceva®) Treatment in Patients With Locally Advanced or Metastatic Non-small Cell Lung Cancer Who Present Activating Mutations in the Tyrosine Kinase Domain of the Epidermal Growth Factor Receptor
Brief Title: A Study of Tarceva (Erlotinib) in Patients With Locally Advanced or Metastatic Non-small Cell Lung Cancer Who Present EGFR Mutations
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML25575
Record Dates: First submitted 2011-01-24; First posted 2011-02-01 (Estimated); Results first posted 2015-06-02 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-05

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: erlotinib [Tarceva]

INTERVENTIONS:
Drug: erlotinib [Tarceva] — 150 mg daily orally

SUMMARY:
This single arm, open-label study will assess the efficacy and safety of Tarceva (erlotinib) in patients with locally advanced or metastatic non-small cell lung cancer with epidermal growth factor receptor (EGFR) mutations. Patients will receive Tarceva at a dose of 150 mg daily orally until disease progression or unacceptable toxicity occurs.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/=18 years of age
* Locally advanced or metastatic (stage III/IV) non-small cell lung cancer with EGFR mutations
* Measurable disease according to RECIST criteria
* ECOG performance status 0-2
* Adequate haematological, renal and liver function

Exclusion Criteria:

* Previous chemotherapy or therapy against EGFR for metastatic disease
* History of another malignancy, except for in situ carcinoma of the cervix, adequately treated basal cell skin carcinoma, or radically treated prostate carcinoma with good prognosis
* Symptomatic cerebral metastases
* Pre-existing parenchymal lung disease such as pulmonary fibrosis
* Concomitant use of coumarins

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-10; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (5):
- Finland (5):
  - Helsinki
  - Kuopio
  - Oulu
  - Pori
  - Turku

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants underwent EGFR mutation testing at Screening. Those positive for the EGFR mutation and who met eligibility criteria (number of participants [n] = 3) received treatment with erlotinib. The remaining participants (n = 21) were followed for overall survival but did not receive treatment.
Groups:
- Erlotinib: Participants positive for the epidermal growth factor receptor (EGFR) mutation and who met eligibility criteria received treatment with erlotinib, 150 milligrams (mg) orally once daily until disease progression or unacceptable toxicity.
- Untreated: Participants without the EGFR mutation were followed for overall survival but did not receive treatment. Additionally, participants positive for the EGFR mutation who were excluded from treatment were followed for overall survival.
Period: Overall Study
Arm/Group | Erlotinib | Untreated
Started | 3 | 21
Completed | 0 | 0
Not Completed | 3 | 21
Not completed — Death | 2 | 12
Not completed — Lost to Follow-up | 1 | 6
Not completed — Protocol Violation | 0 | 3

BASELINE CHARACTERISTICS:
Population: All erlotinib-treated participants who received at least one dose of erlotinib, in addition to all enrolled untreated patients, were included in the analysis.
Groups:
- Erlotinib: Participants positive for the EGFR mutation and who met eligibility criteria received treatment with erlotinib, 150 mg orally once daily until disease progression or unacceptable toxicity.
- Untreated: Participants without the EGFR mutation were followed for overall survival but did not undergo treatment. Additionally, participants positive for the EGFR mutation who were excluded from treatment were followed for overall survival.
- Total: Total of all reporting groups
Arm/Group | Erlotinib | Untreated | Total
Number analyzed (Participants) | 3 | 21 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 75 (7.6) | 67 (8.4) | 68 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 13 | 15
  Male | 1 | 8 | 9

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) Among Erlotinib-Treated Participants With the EGFR Mutation
Description: PFS was defined as the time from the first dose of erlotinib to the first documentation of disease progression or death, whichever occurred first. Tumor progression was determined using Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1), which defines progression as a 20 percent (%) or greater increase in the sum of diameters of target lesions with an absolute increase of at least 5 millimeters (mm), or the appearance of one or more new lesions. PFS was calculated in months as [first event date minus first dose date plus 1] divided by 30.44.
Time Frame: Per standard of care (every 3 months) until discontinuation for up to approximately 2 years
Population: All Participants Treated: All participants who received at least one dose of erlotinib were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib
Number analyzed (Participants) | 3
months | 13.7 [2.0 to NA] — Data for 1 of 3 participants were censored, and thus a confidence interval upper limit was not reached.

2. Secondary Outcome: Number of Erlotinib-Treated Participants With the EGFR Mutation With an Objective Response Per RECIST v1.1
Description: Objective tumor response was assessed by the investigator using RECIST v1.1 and recorded as complete response (CR), partial response (PR), or unmeasurable. RECIST v1.1 defines CR as disappearance of all target lesions, with short-axis reduction to less than (<) 10 mm for any pathological lymph nodes, and PR as a 30% or greater reduction from baseline in the sum of diameters of target lesions.
Time Frame: Per standard of care (every 3 months) until discontinuation for up to approximately 2 years
Population: All Participants Treated
Measure: Number; unit: participants
Arm/Group | Erlotinib
Number analyzed (Participants) | 3
participants
  Partial response | 2
  Unmeasurable | 1

3. Secondary Outcome: Overall Survival (OS) Among Erlotinib-Treated and Untreated Participants
Description: OS was defined as the time from recorded diagnosis to death from any cause or last patient last visit. OS was calculated in months as [death date or last-known alive date minus diagnosis date plus 1] divided by 30.44.
Time Frame: Per standard of care (every 3 months) until discontinuation for up to approximately 2 years
Population: All Participants Enrolled: All erlotinib-treated participants who received at least one dose of erlotinib, in addition to all enrolled untreated participants, were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib | Untreated
Number analyzed (Participants) | 3 | 21
months | 17.8 [17.6 to NA] — Data for 1 of 3 participants were censored, and thus a confidence interval upper limit was not reached. | 11.3 [8.4 to 11.4]

4. Secondary Outcome: Percentage of Participants Alive at 6 and 12 Months
Description: Death from any cause was documented at 6 and 12 months from recorded diagnosis. The percentage of participants alive at each timepoint was calculated as [number of participants alive divided by number enrolled] multiplied by 100.
Time Frame: At 6 and 12 months
Population: All Participants Enrolled
Measure: Number; unit: percentage of participants
Arm/Group | Erlotinib | Untreated
Number analyzed (Participants) | 3 | 21
percentage of participants
  At 6 months | 100 | 67
  At 12 months | 100 | 24

5. Secondary Outcome: Percentage of Participants With EGFR Mutation at Screening
Description: Participants were tested at Screening for the presence of activating mutations in the tyrosine kinase domain of EGFR. The percentage of participants with mutation was calculated as [number of mutation-positive participants divided by number tested] multiplied by 100.
Time Frame: Screening
Population: All Participants Enrolled
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- All Participants: All participants underwent EGFR mutation testing at Screening. Those positive for the EGFR mutation and who met eligibility criteria (n = 3) received treatment with erlotinib, 150 mg orally once daily until disease progression or unacceptable toxicity. The remaining participants (n = 21) were followed for overall survival but did not receive treatment.
Arm/Group | All Participants
Number analyzed (Participants) | 24
percentage of participants | 17 [2 to 32]

ADVERSE EVENTS:
Time Frame: Up to 2 years
Description: Only participants treated with erlotinib were assessed for adverse events.
Arm/Group | Erlotinib
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib (N=3)
Epidural catheter infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib (N=3)
Alopecia (Skin and subcutaneous tissue disorders) | 1
Bleeding from mouth (Gastrointestinal disorders) | 1
Eye infection (Infections and infestations) | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Periosteal reaction (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Paraparesis (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.